CLINICAL TRIAL: NCT02720159
Title: A Prospective, Early Feasibility Study to Characterize the Efficacy and Safety of a Percutaneous Osseointegrated Prosthesis
Brief Title: Early Feasibility Study of the Percutaneous Osseointegrated Prosthesis (POP)
Acronym: POP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POP
Record Dates: First submitted 2016-03-08; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Amputee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TREATMENT (Experimental)
  Interventions: Device: Percutaneous Osseintegrated Prosthesis

INTERVENTIONS:
Device: Percutaneous Osseintegrated Prosthesis

SUMMARY:
The purpose of the clinical study is to characterize the efficacy and safety of a Percutaneous Osseointegrated Prosthesis (POP) device that can provide a satisfactory platform for direct skeletal attachment of prosthetic limbs, which includes a subdermal seal, thus allowing a proper biobarrier around the implant.

ELIGIBILITY:
Inclusion Criteria:

* US Military veteran with transfemoral amputation that is not a result of dysvascular disease
* Has used or is using a "socket suspension technology" prosthesis
* Use of non-propulsive, passive microprocessor-regulated devices
* Agrees not to participate in high levels of physical activity while in the study
* Subject meets anatomical and eligibility criteria for the investigational device

Exclusion Criteria:

* Currently on active military duty
* More than 1 limb amputated
* Has insulin dependent or adult onset diabetes
* Recent tobacco use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Assess AP & Lateral x-rays for osteolysis, radioulucencies indicative of component moevent and orientation and stress shielding or bone remodeling around the implant | 1 year
Changes in Bone Mineral Density as collected using DEXA scan | 1 year
Changes in implant exit site using Modified Holgers Skin Metric | 1 yr
Analyze measurable changes in the stoma punch | 1 year
Analyze changes of walking and standing | 1 year
  Three dimensional motion capture of walking and standing through a calibration volume that contains force plates
Analyze changes in metabolic efficiency | 1 year
  Measure CO2 and O2 exhaled, total energy cost for walking at slow, normal, fast; self-selected and/or fixed speeds while wearing a two-way valve.
Analyze changes in 6 minute walk test | 1 year
Assess changes in Donning and Doffing prosthetic time | 1 year
Assess changes in Comprehensive High-Level Activity Mobility Predictor (CHAMP) test | 1 year
Changes in psychosocial adjustment with the Trinity Amputation and Prosthesis Experience Scales - Revised (TAPES-R) Part I, 37 questions | 1 yr
Changes in depressive symptomatology using the Center for Epidemiologic Studies Depression Scale Revisited (CES-D) | 1 yr
Changes in consequences of pain on relevant aspects of persons' lives using PROMIS: Pain Interference questions | 1 yr
Changes in ability to carry out activities that require physical actions using PROMIS: Physical Function | 1 yr
Changes in overall quality of life using QOL Visual Analog Scale, no numerical weighting | 1 yr
Changes in at-home prosthetic usage using StepWatch activity monitor | 1 yr

CONTACTS AND LOCATIONS:
Locations (1):
- George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Sinclair S, Beck JP, Webster J, Agarwal J, Gillespie B, Stevens P, Gililland J, Kubiak E. The First FDA Approved Early Feasibility Study of a Novel Percutaneous Bone Anchored Prosthesis for Transfemoral Amputees: A Prospective 1-year Follow-up Cohort Study. Arch Phys Med Rehabil. 2022 Nov;103(11):2092-2104. doi: 10.1016/j.apmr.2022.06.008. Epub 2022 Jul 29. PMID 35908658